CLINICAL TRIAL: NCT03471650
Title: A Phase II Study to Evaluate the Performance of PSMA-targeted 18F-DCFPyL PET/CT for the Detection of Clinically Significant Prostate Cancer in Men With an Elevated PSA
Brief Title: Study of PSMA-targeted 18F-DCFPyL PET/CT for the Detection of Clinically Significant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J17149; IRB00139990 (Other: JHMIRB)
Record Dates: First submitted 2018-03-02; First posted 2018-03-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: J17149; PSMA; 18F-DCFPyL PET/CT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL Injection (Experimental): A bolus of ~9 mCi (333 MBq) of 18F-DCFPyL will be injected by slow IV push.
  Interventions: Drug: 18F-DCFPyL Injection

INTERVENTIONS:
Drug: 18F-DCFPyL Injection — A bolus of ~9 mCi (333 MBq) of 18F-DCFPyL will be injected by slow IV push.
  Other Names: PyL

SUMMARY:
This is a phase II, single-center, open-label, trial to evaluate the diagnostic accuracy of PSMA-targeted 18F-DCFPyL PET/CT for detecting clinically significant prostate cancer in a screening population.

DETAILED DESCRIPTION:
This is a phase II, single-center, open-label, trial to evaluate the diagnostic accuracy of PSMA-targeted 18F-DCFPyL PET/CT for detecting clinically significant prostate cancer in a screening population. 150 biopsy-naïve patients with an elevated PSA (2-10 ng/mL) will be enrolled in this study.

Within 28 days of informed consent, patients will undergo an 18F-DCFPyL PET/CT. All scans will be read by a single experienced radiologist who will identify regions of interest (ROI) with discrete radiotracer uptake. The maximum SUV value (SUVmax) of each ROI will be recorded. For patients without a detectable ROI, the mean SUV (SUVmean) of a 1-2 cm volume of the prostate will instead be recorded.

One to 28 days following PET/CT imaging, a systematic 12 to 14 core TRUS-guided prostate biopsy will be performed. Immediately following completion of systematic TRUS biopsies, fusion-targeted biopsies of all PET and/or MRI visible lesions will be performed, taking an additional 2 to 3 cores from each radiographic ROI. All biopsy cores will be assessed for Gleason score and percent cancer involvement.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* PSA of 2-10 ng/mL
* Clinical stage T1c-T2a on digital rectal exam
* Elect to undergo TRUS-guided prostate biopsy as part of routine clinical care
* Willingness to sign informed consent and comply with all protocol requirements

Exclusion Criteria:

* History of prior prostate biopsy
* Administered a radioisotope ≤5 physical half-lives prior to the date of study PET/CT
* Administered IV X-ray contrast medium ≤24 hours prior to the date of study PET/CT
* Administered oral contrast medium ≤120 hours prior to the date of study PET/CT
* Any medical condition or other circumstances that in the opinion of the investigators compromise obtaining reliable data or achieving the study objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is For Prostate Cancer in Men
Enrollment: 150 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2027-03-07 (Estimated); Study Completion 2027-03-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 18F-DCFPyL PET/CT to detect clinically significant prostate cancer on prostate biopsy relative to serum prostate specific antigen (PSA) | 4 years
  Measure the diagnostic accuracy of 18F-DCFPyL PET/CT and compare it with serum PSA for detecting clinically significant prostate cancer on prostate biopsy

SECONDARY OUTCOMES:
Sensitivity of 18F-DCFPyL PET/CT relative to PSA | 4 years
  Measure the diagnostic accuracy of 18F-DCFPyL PET/CT relative to serum PSA for detecting clinically significant prostate cancer as defined by the following alternative definitions: Gleason score ≥4+3=7; Gleason score ≥3+4 or >50% involvement of ≥1 core with Gleason score ≥3+3=6 prostate cancer; Gleason score ≥3+4 or >70% involvement of ≥1 core with Gleason score ≥3+3=6 prostate cancer; Gleason score ≥3+4=7, or >2 cores with Gleason score ≥3+3=6, or >50% involvement of ≥1 core with Gleason score ≥3+3=6 prostate cancer.
Sensitivity of 18F-DCFPyL PET/CT for detecting clinically significant prostate cancer relative to mpMRI | 4 years
  Measure the diagnostic accuracy of 18F-DCFPyL PET/CT relative to mpMRI for detecting clinically significant prostate cancer by the various tested definitions
Sensitivity and diagnostic accuracy of 18F-DCFPyL PET/CT relative to the phi blood test for detecting clinically significant prostate cancer by the various tested definitions | 4 years
  Measure the diagnostic accuracy of 18F-DCFPyL PET/CT relative to the phi blood test for detecting clinically significant prostate cancer by the various tested definitions

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Allaf, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- SKCCC, Baltimore, Maryland, United States